CLINICAL TRIAL: NCT04371627
Title: Viaskin® Peanut (DBV712) Expanded Access Protocol in Peanut-Allergic Children
Brief Title: Viaskin® Peanut (DBV712) Expanded Access Protocol
Status: No longer available | Type: Expanded Access
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: V712-EAP01
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Peanut Allergy
Keywords: Peanut allergy; EPIT; Epicutaneous; Immunotherapy; Viaskin®
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Viaskin Peanut — Daily epicutaneous delivery
  Other Names: DBV712

SUMMARY:
This is an open label expanded access program for male and female patients ≥ 4 years old.

DETAILED DESCRIPTION:
This study is an open-label Intermediate-size EAP designed to provide treatment access for eligible Peanut-Allergic Children. This EAP entails visits every three months to assess patient status, safety, and to provide drug supply. Viaskin® Peanut treatment will continue until, in the clinical judgment of the Investigator, the patient is no longer benefiting from continuation of the treatment, the drug becomes approved and available by prescription, or the study is terminated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 4 years of age
* Prior participation in a Viaskin® Peanut REALISE or PEOPLE clinical study for peanut-allergic patients

Exclusion Criteria:

* Pregnancy or lactation or planning a pregnancy.
* Generalized dermatologic disease (for example, active atopic dermatitis, uncontrolled generalized active eczema, ichthyosis vulgaris) extending widely on the skin and especially on the back with no intact zones to apply the Viaskin® patches.
* Patients who developed hypersensitivity to excipients of the Viaskin® patches.
* Received or planning to receive anti-tumor necrosis factor drugs or anti-IgE drugs (such as omalizumab) or any biologic immunomodulatory therapy.
* Receiving or planning to receive any other type of immunotherapy to any food (for example, EPIT, OIT, or SLIT or specific oral tolerance induction) or any aeroallergen or venom immunotherapy during their participation in the study.
* Use of cyclosporine or other immunosuppressive agents within 3 months before entering the study. Topical calcineurin inhibitors are permitted.
* A history of important non-compliance during the REALISE or PEOPLE studies. Important non-compliance includes patients not applying the patches for 60 or more days in total and/or for 30 or more consecutive days during the REALISE or PEOPLE studies.

Ages: 4 Years to 12 Years | Sex: All
Age Groups: Child